CLINICAL TRIAL: NCT01722136
Title: We Walk - Energy Expenditure and Health Outcomes in Older, Sedentary Women.
Brief Title: "We Walk": Impact of Exercise Dose on Health Outcomes Among Women Ages 60-75
Acronym: WW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Xuewen Wang, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00016306
Record Dates: First submitted 2012-10-24; First posted 2012-11-06 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2016-05

CONDITIONS: Condition
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dosage (Experimental): Exercise dose of 8kcal/kg/week
  Interventions: Behavioral: Low Dosage
- High Dosage (Experimental): Exercise dose 14kcal/kg/week
  Interventions: Behavioral: High Dosage

INTERVENTIONS:
Behavioral: Low Dosage — Exercise dose of 8kcal/kg/week
  Arms: Low Dosage
Behavioral: High Dosage — Exercise dose of 14kcal/kg/week
  Arms: High Dosage

SUMMARY:
The overall goal is to determine whether any energy expenditure compensation in response to 16 weeks of aerobic exercise at a higher-dose is greater compared to a lower-dose intervention in older women, and to begin to investigate underlying physiological mechanisms that influence energy expenditure changes in older women.

DETAILED DESCRIPTION:
The overall goal is to determine whether any energy expenditure compensation in response to 16 weeks of aerobic exercise at a higher-dose is greater compared to a lower-dose intervention in older women, and to begin to investigate underlying physiological mechanisms that influence energy expenditure changes in older women. Changes in all components of energy expenditure, as well as concentrations of plasma leptin and serum free T3, in response to the two different exercise programs (14 and 8 kcal/kg body weight weekly, 60-65% VO2max, 4 days/wk) will be compared in older, non-obese women (60-75 yrs, BMI=18-30 kg/m2).

Specific Aim 1: To determine whether differential changes in total daily energy expenditure and its components occur in older women in response to two exercise programs of different doses. State-of-the-art methods will be used (total daily energy expenditure by doubly labeled water; non-exercise activity thermogenesis using Physical Activity Monitoring System; resting metabolic rate and thermic effect of food via indirect calorimetry).

Primary Hypothesis: Due to a greater decline in NEAT, women will exhibit a smaller increase in total daily energy expenditure in response to the higher-dose, compared to the lower-dose, exercise program, despite greater increases in resting metabolic rate and thermic effect of food.

Specific Aim 2: To explore whether differential changes occur in plasma leptin and serum free triiodo-L-thyronine (free T3) concentrations in older women in response to 16-week aerobic exercise programs of two different doses.

We hypothesize that in response to the higher-dose exercise program, women will exhibit larger decreases in plasma leptin and serum free T3 concentrations, compared to the lower-dose exercise program.

We will also determine whether women exhibit greater improvements in plasma lipids, insulin sensitivity (using homeostasis model assessment, HOMA, score), blood pressure, and aerobic fitness in response to the higher-dose, compared to the lower-dose, exercise program.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30
* Sedentary (exercising less than 20 minutes no more than 3 times per week)
* Non-smoking
* Weight stable (+/- 5%) over past 3 months

Exclusion Criteria:

* Self-reported cardiovascular disease
* Additional self-reported medical conditions
* Medications known to affect metabolism
* Excess caffeine use
* Self-reported contradictions according to ACSM
* Unwillingness to provide informed consent

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline total daily energy expenditure and its components (resting metabolic rate, thermic effect of food, non-exercise activity thermogenesis)in 4 months | Baseline (pre-intervention); 4 months (post-intervention)

SECONDARY OUTCOMES:
Change from baseline plasma leptin and serum free triiodo-L-thyronine (free T3) concentrations in 4 months | Baseline (pre-intervention); 4 month (post-intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Xuewen Wang, PhD, MEd, BM, Principal Investigator — University of South Carolina
Locations (1):
- Public Health Research Center University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- See also: Brief description of study for potential participants — http://wewalk.sc.edu